CLINICAL TRIAL: NCT05283616
Title: A Randomized Controlled Study Comparing Different Doses of Pegfilgrastim as Support for Adjuvant Chemotherapy for Breast Cancer
Brief Title: Reduced Dose of Pegfilgrastim as Support for Chemotherapy for Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-CS-003
Record Dates: First submitted 2022-03-02; First posted 2022-03-17 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Neutropenia
MeSH Terms: conditions — Neutropenia | interventions — pegfilgrastim

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pegfilgrastim 3mg (Experimental): Pegfilgrastim 3mg per chemotherapy cycle
  Interventions: Drug: Pegfilgrastim
- pegfilgrastim 6mg (Active Comparator): Pegfilgrastim 6mg per chemotherapy cycle
  Interventions: Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Pegfilgrastim — Pegfilgrastim 3mg per chemotherapy cycle

SUMMARY:
Pegfilgrastim is a long-acting recombinant human granulocyte-colony stimulating factor as support for chemotherapy, which can be used conveniently.

According to the package inserts in America, Europe, and China, the recommended dose for pegfilgrastim is 6mg per cycle, while it is recommended at a dose of 3.6mg in Japan. It is still unclear whether pegfilgrastim 3mg can produce similar efficacy with pegfilgrastim 6mg.

In this trial, the investigators prospectively compared the efficacy and safety of pegfilgrastim 3mg with 6mg in patients with breast cancer receiving AC regimen, a commonly used regimen in adjuvant chemotherapy for breast cancer.

DETAILED DESCRIPTION:
All patients received AC regimen (epirubicin or pirarubincin in combination with cyclophosphamide) intravenously. Epirubicin 90mg/m^2 (or pirarubicin 60mg/m^2) and cyclophosphamide 600mg/m^2 were administered on day 1 of the chemotherapy cycle. AC regimen was administered bi-weekly or 3-weekly.

Eligible patients were randomly assigned to 3mg arm (the study arm) and 6mg arm (the control arm) in a 1:1 ratio, stratified according to body weight (≤60kg or >60kg). Patients in the study arm and the control arm received a subcutaneous injection of 3mg PEG-rhG-CSF and 6mg, respectively, forty-eight hours after completing chemotherapy infusion.

ELIGIBILITY:
Inclusion Criteria:

* female aged 18-69 years
* diagnosed pathologically as early breast cancer
* with indication for adjuvant chemotherapy and suitable for AC regimen (epirubicin and cyclophosphamide, or pirarubicin and cyclophosphamide, planned chemotherapy with taxanes after AC regimen were allowed)
* received no prior chemotherapy (chemotherapy naïve)
* have Karnofsky performance status ≥ 80,
* baseline hemoglobin ≥90g/L, white blood cell count ≥4.0X10^9/L,ANC≥2.0X10^9/L, platelet count ≥100X10^9
* adequate cardiac, hepatic and renal function

Exclusion Criteria:

* enrolled onto or had not yet completed other investigational drug trials
* allergic to any component of PEG-rhG-CSF injection, or other biological products derived from genetically engineering Escherichia coli;
* pregnant or lactating women;
* previous large volume radiotherapy, or prior bone marrow or stem-cell transplantation

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
timely recovery of ANC | 1 month
  The proportion of patients with absolute neutrophil count (ANC) ≥2.0×10^9/L before the second chemotherapy cycle. Blood routine test was used.

SECONDARY OUTCOMES:
febrile neutropenia in cycle1 | 1 month
  the incidence of neutropenia with fever in cycle 1. Blood test was used and body temperature was taken.
grade 3/4 neutropenia in cycle 1 | 1 month
  the incidence of absolute neutrophil count (ANC) <1.0×10^9/L before the second chemotherapy cycle. Blood routine test was used.
grade 4 neutropenia in cycle 1 | 1 month
  the incidence of absolute neutrophil count (ANC) <0.5×10^9/L before the second chemotherapy cycle. Blood routine test was used.
hospitalization due to neutropenia | 1 month
  the incidence of unplanned hospitalization due to neutropenia

OTHER OUTCOMES:
adverse events | 1 month
  the profile and incidence of adverse events. Symptoms and signs were observed; blood routine test and blood biochemistry tests were performed.

CONTACTS AND LOCATIONS:
Overall Officials: Pin Zhang, Principal Investigator — Department of Medical Oncology, Cancer Hospital, CAMS
Locations (1):
- Department of Medical Oncology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No